CLINICAL TRIAL: NCT05771974
Title: A Randomized Controlled Trial Using Surgical Gloves to Prevent Chemotherapy-induced Peripheral Neuropathy by Paclitaxel in Breast Cancer Patients
Brief Title: The AIUR Trial: Surgical Gloves to Prevent Peripheral Neuropathy
Acronym: AIUR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Young-Joon Kang (Other)
Responsible Party: Sponsor-Investigator, Young-Joon Kang, Assistant Professor, Incheon St.Mary's Hospital
Organization: Incheon St.Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AIUR trial
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compression therapy using surgical gloves (Experimental): Study participants wear two-layer of normal-sized surgical gloves on both hands during chemotherapy infusion
  Interventions: Device: Compression therapy using surgical gloves
- Control (No Intervention): No intervention is provided on both hands.

INTERVENTIONS:
Device: Compression therapy using surgical gloves — Intervention group wear two-layer of normal-sized surgical gloves on both hands during chemotherapy infusion
  Arms: Compression therapy using surgical gloves

SUMMARY:
This study aims to demonstrate the preventive effect of compression therapy using surgical gloves in chemotherapy-induced peripheral neuropathy. Patient-reported outcome measures (PROMs) are utilized for comparing the change in neuropathic pain between intervention and control groups. Among the PROMs, the neurotoxicity component of the functional Assessment of Cancer Therapy-taxane (FACT-Tax) is used for good and poor outcomes between baseline and post-chemotherapy in paclitaxel-treated breast cancer patients.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) is associated with side effects of taxanes, including paclitaxel. The common side effect may adversely affect the quality of life. However, no treatment for CIPN can be strongly recommended. Therefore, prevention is important. Cryotherapy, compression therapy, and exercise therapy can be considered for prevention, but no definitive recommendations are available. Studies with wider sample sizes are needed to confirm the efficacy and the preventive methods are complex for application. The study use surgical gloves for compression therapy to reduce discomfort and increase compliance with the procedure.

Patients with stage II-III breast cancer who receive paclitaxel chemotherapy for at least 12 weeks in six academic hospitals in South Korea will participate in the study. The study design is a multicenter, open-label, randomized controlled trial. The patients are randomly assigned to intervention or control groups. Intervention patients will wear two-layer of normal-sized surgical gloves on both hands during chemotherapy infusion. The primary outcome is to demonstrate the preventive effect of compression therapy using surgical gloves as measured by the change in the neurotoxicity of FACT-Tax questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 19 years, under 70 years old
* Stage II-III breast cancer
* No distant metastasis
* Patient scheduled to be receiving adjuvant or neoadjuvant paclitaxel for at least 12 weeks
* Signed informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥60%)

Exclusion Criteria:

* Recurred breast cancer
* Patients who have previously received treatment that could cause neuropathy; taxane or platinum-based chemotherapy, antitubulins, proteasome inhibitors
* Known history of neuropathy
* Chronic kidney disease
* Raynaud's phenomenon
* Peripheral vascular disease; peripheral arterial ischemia
* Cold intolerance
* Allergy in natural rubber latex or surgical gloves
* Patients who have dermatitis, wound, or musculoskeletal problems in hand at enrollment
* Current use medications which may mitigate chemotherapy-induced peripheral neuropathy; duloxetine, gabapentin/pregabalin, Baclofen-amitriptyline-ketamine (BAK; topical amitriptyline, ketamine, ±baclofen), oral cannabinoids, tricyclic antidepressants, ganglioside-monosialic acid

Ages: 19 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the 11 items neurotoxicity component of the Functional Assessment of Cancer Therapy-Taxane (FACT-NTX) Therapy subscale | Before starting paclitaxel course (baseline), and 1~2 weeks from finishing paclitaxel course chemotherapy (target)
  The change in FACT-NTX will be divided into a good outcome (change in FACT-NTX less than five from baseline to target timeframe) versus a poor outcome (change in FACT NTX greater than or equal to five from baseline to target timeframe). The difference in the number of poor outcome participants will compare between the two groups. The FACT-NTX is 5-point Likert-type scale. Each item measures on a 0-4 scale (0, not at all; 4, very much). A greater change in the FACT-NTX score was considered a clinically meaningful increase in CIPN.

SECONDARY OUTCOMES:
Changes in 16 items component of the Functional Assessment of Cancer Therapy-Taxane (FACT-Taxane) Therapy subscale | Baseline, during paclitaxel course (about 1.5 months after starting), 1~2 weeks from finishing course, and six months after finishing paclitaxel course
  The score changes in 16 items (neurotoxicity and taxane) component of the FACT-Taxane scale will be compared between the two groups. The FACT-Taxane is 5-point Likert-type scale. Each item measures on a 0-4 scale (0, not at all; 4, very much). A scale of 0 indicates a better outcome, and 4 indicates a worse outcome.
Changes in 27 items component of the Functional Assessment of Cancer Therapy-General (FACT-G) scale | Baseline, during paclitaxel course (about 1.5 months after starting), 1~2 weeks from finishing course, and six months after finishing paclitaxel course
  The score changes in general 27 items component of the FACT-G scale will be compared between the two groups. The FACT-G consists of four well-being subscales; physical well-being (7-item), social/family well-being (7-item), emotional well-being (6-item), and functional well-being (7-item). The FACT-G is 5-point Likert-type scale (0, not at all; 4, very much). For physical and emotional well-being, the higher the sum of scores, the lower the quality of life; for social/family and functional well-being, the higher the sum of scores, the higher the quality of life.
Changes in the 11 items neurotoxicity component of the Functional Assessment of Cancer Therapy-Taxane (FACT-NTX) Therapy subscale at additional periods. | During paclitaxel course (about 1.5 months after starting) and six months after finishing paclitaxel course
  The change in FACT-NTX will be divided into a good outcome (change in FACT-NTX less than five from baseline to target timeframe) versus a poor outcome (change in FACT NTX greater than or equal to five from baseline to target timeframe). The difference in the number of poor outcome participants will compare between the two groups. The FACT-NTX is 5-point Likert-type scale. Each item measures on a 0-4 scale (0, not at all; 4, very much). A greater change in the FACT-NTX score was considered a clinically meaningful increase in CIPN.
Change in National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) for CIPN | Baseline, during paclitaxel course (about 1.5 months after starting), 1~2 weeks from finishing course, and six months after finishing paclitaxel course
  NCI-CTCAE for CIPN is a method for reporting adverse event severity by a combination of clinical evaluation. The adverse effects of CIPN to be investigated are peripheral motor, sensory neuropathy, dysesthesia, paresthesia, neuralgia, and skin/nail toxicity.
Comfort with intervention scale score | during paclitaxel course (about 1.5 months after starting), 1~2 weeks from finishing course, and six months after finishing paclitaxel course
  Comfort with the intervention (two-layer of surgical gloves) will be assessed on 4-point scale. The points are classified 0=dissatisfied; 1=not satisfied; 2=satisfied; 3=very satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Incheon St. Mary's Hospital, Incheon, Bupyeong, South Korea

REFERENCES:
- [Background] Kang YJ, Yoon CI, Yang YJ, Baek JM, Kim YS, Jeon YW, Rhu J, Yi JP, Kim D, Oh SJ. A randomized controlled trial using surgical gloves to prevent chemotherapy-induced peripheral neuropathy by paclitaxel in breast cancer patients (AIUR trial). BMC Cancer. 2023 Jun 20;23(1):570. doi: 10.1186/s12885-023-11079-8. PMID 37340369